CLINICAL TRIAL: NCT00745745
Title: Septal Positioning of Ventricular ICD Leads
Brief Title: Septal Positioning of Ventricular Implanted Cardioverter Defibrillator (ICD) Leads
Acronym: SPICE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: T83
Record Dates: First submitted 2008-09-02; First posted 2008-09-03 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Ventricular Tachycardia; Ventricular Fibrillation
MeSH Terms: conditions — Tachycardia, Ventricular; Ventricular Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Apical ICD lead placement
  Interventions: Device: Device Implantation
- 2 (Experimental): Mid-Septal ICD lead placement
  Interventions: Device: Device Implantation

INTERVENTIONS:
Device: Device Implantation — ICD lead implantation
  Other Names: CE marked ICD/CRT-D from St. Jude Medical and compatible CE marked ICD- and; pacemaker- and active fixation ICD-leads

SUMMARY:
This clinical trial is a multi center, prospective, randomized, parallel study designed to compare septal to apical ICD lead placement.

DETAILED DESCRIPTION:
The primary objective of this clinical investigation is to demonstrate that septal positioning of the right ventricular defibrillation lead is not inferior to the apical positioning in terms of safety and efficacy in a population of ICD recipients.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 years
* Signed written informed consent
* Approved indication for implantation of ICD / CRT-D device

Exclusion Criteria:

* Preexisting transvenous RV pacemaker or ICD leads
* Pacemaker dependency without sufficient intrinsic rhythm (≤ 30min-1)
* Hypertrophic obstructive cardiomyopathy
* Presence of intra-aortic balloon pump
* Inotropic drug (not digitalis) necessary for hemodynamic support
* Inability to perform VF induction testing due to anticipated high risk
* Condition likely to limit cooperation
* Unable to give informed consent
* Pregnancy or planned pregnancy in the next 6 months
* Patients with planned cardiac surgery within the next 3 months following randomization
* Patient is currently participating in a clinical investigation that includes an active treatment arm.
* Acute myocardial infarction within the previous 4 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 299 (Actual)
Dates: Start 2008-08; Primary Completion 2011-06 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Event free survival of RV-ICD-lead related complications | 3 months after implantation

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Kolb, MD, Principal Investigator — Deutsches Herzzentrum München des Freistaates Bayern
Locations (21):
- Germany (20):
  - Ost-Alb Klinikum, Aalen
  - SLK-Kliniken Heilbronn GmbH Klinikum am Plattenwald, Bad Friedrichshall
  - Segeberger Kliniken GmbH, Bad Segeberg
  - Städtisches Klinikum Brandenburg, Brandenburg
  - Medizinisches Versorgungszentrum, Dachau
  - Krankenhaus Düren gGmbH Akademisches Lehrkrankenhaus der RWTH-Aachen, Düren
  - Klinikum Esslingen, Esslingen am Neckar
  - Universitätsklinik Freiburg, Freiburg im Breisgau
  - Herzkatheterlabor der Kardiologischen Praxis am Krankenhaus Neu-Bethlehem gGmbH, Göttingen
  - Asklepios Klinik St. Georg, Hamburg
  - Oberhavel Kliniken GmbH Klinik Hennigsdorf, Hennigsdorf
  - Krankenhaus Landshut-Achdorf, Landshut
  - Universitätsklinikum Leipzig AÖR, Leipzig
  - Kliniken Ludwigsburg-Bietigheim, Ludwigsburg
  - Märkische Kliniken GmbH Klinikum Lüdenscheid, Lüdenscheid
  - Klinikum Mannheim gGmbH Fakultät für Klinische Medizin Mannheim der Universität Heidelberg, Mannheim
  - Maria-Hilf Franziskus-Krankenhaus, Mönchengladbach
  - Deutsches Herzzentrum Muenchen, Munich
  - Niels-Stensen-Kliniken Marienhospital Osnabrück, Osnabrück
  - Klinkum Peine gGmbH, Peine
- Henry Dunant Hospital, Athens, Greece

REFERENCES:
- [Derived] Kolb C, Solzbach U, Biermann J, Semmler V, Kloppe A, Klein N, Lennerz C, Szendey I, Andrikopoulos G, Tzeis S, Asbach S; SPICE-investigators. Safety of mid-septal electrode placement in implantable cardioverter defibrillator recipients--results of the SPICE (Septal Positioning of ventricular ICD Electrodes) study. Int J Cardiol. 2014 Jul 1;174(3):713-20. doi: 10.1016/j.ijcard.2014.04.229. Epub 2014 Apr 26. PMID 24838056